CLINICAL TRIAL: NCT01556581
Title: Effectiveness and Subsequent Healthcare Use Associated With Early Physical Therapy Access Compared With a Stepped Usual Care Approach for Treatment of Low Back Pain.
Brief Title: Comparative Effectiveness of Early Physical Therapy Versus Usual Care for Low Back Pain
Acronym: COMPETE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Madigan Army Medical Center (U.S. Federal Agency)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency); William Beaumont Army Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 211107
Record Dates: First submitted 2012-03-14; First posted 2012-03-16 (Estimated); Results first posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-06

CONDITIONS: Low Back Pain
Keywords: back pain; primary care; physical therapy
MeSH Terms: conditions — Low Back Pain; Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (UC) (Active Comparator): The usual care (UC) group will be managed with stepped care approach, receiving a screening exam, advice, education, activity limitation profile and medications if needed, but no early physical therapy.
  Interventions: Procedure: Usual Care (UC)
- Early Physical Therapy (PT) (Active Comparator): All subjects in this group will get usual care approach in addition to immediately receiving eight sessions of physical therapy based on a pragmatic treatment based classification system for treating low back pain.
  Interventions: Procedure: Early Physical Therapy (PT)

INTERVENTIONS:
Procedure: Usual Care (UC) — Initial management for all patients will include an activity-limiting profile for up to 30 days and a 10-day supply of medications if needed (NSAIDs and muscle relaxers). All patients will then receive advice and education about the favorable natural history of LBP and the advantages of remaining as active as possible. All patients will be recommended to follow-up with their primary care provider using normal procedures if they are not satisfied with their progress.
  Arms: Usual Care (UC)
Procedure: Early Physical Therapy (PT) — Patients in the early PT group will receive the same treatment as the usual care group, but will then be referred to physical therapy within 3 days. The physical therapy treatment will be based on the Treatment Based Classification system (an approach that places patients into either an extension-oriented, core strength/stabilization, or a spinal manipulation treatment group based on signs and symptoms).
  Arms: Early Physical Therapy (PT)

SUMMARY:
The primary purpose of this study is to compare the effectiveness of two management strategies for patients with a recent onset of low back pain (LBP). One is based on usual care and the other is based on early access to physical therapy following a pragmatic treatment-based classification approach. The secondary purposes are to compare the subsequent healthcare utilization associated with two management strategies as well as to evaluate the importance of psychosocial factors on outcomes within both groups of treatment. The overall hypothesis guiding the study is that the additional initial treatment expense incurred by early implementation will result in superior short-term clinical effectiveness, and will be more cost-effective in the long-term due to reduced healthcare utilization. We will also explore the importance of psychosocial factors on outcomes within both treatment groups, which may provide insights for further improving treatment strategies.

DETAILED DESCRIPTION:
The specific aims of this study are the following:

1. Compare the effectiveness of two primary care management strategies for patients with a recent onset of combat-related LBP. We hypothesize early physical therapy access for these Soldiers will result in greater improvements in function and quality of life over 1 year as compared to a stepped care strategy.
2. Compare the subsequent healthcare utilization associated with two management strategies for patients with a recent onset combat-related LBP. We hypothesize early physical therapy access will result in decreased healthcare utilization over 1 year as compared to a stepped care strategy.
3. Evaluate the importance of psychosocial factors on outcomes within both groups of treatment.

ELIGIBILITY:
Inclusion Criteria -

* Military personnel on active duty and eligible for healthcare at a military treatment facility
* A primary complaint of low back pain defined as symptoms of pain and/or numbness between the 12th rib and buttocks with or without symptoms into the leg(s), which, in the opinion of the provider, are originating from tissues of the lumbar region.
* Duration of current episode of low back pain < 90 days
* Age 18 - 60 years (or emancipated minors on active duty)
* Available for the following 4 weeks to complete a regimen of treatment

Exclusion Criteria:

* Oswestry Disability Index < 20%
* History of receiving any medical care for this episode of low back pain within the last 3 months
* Prior surgery to the thoraco-lumbar spine or pelvis
* This episode of back pain is due to a traumatic fracture
* Pending a medical or physical evaluation board or discharge process, pending any litigation related to the condition, or planning on getting out of the military within the next 9 months.
* Any "red flags" that would indicate a potentially serious condition or other significant disease process. These could include but not limited to cauda equina syndrome, large or rapidly progressing neurological deficit, fracture, cancer, ankylosing spondylitis, or other systemic disease.
* Current episode occurred because of a motor vehicle accident
* Currently pregnant (or history of pregnancy in the previous 6 months)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2016-07-27 (Actual); Study Completion 2017-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Fritz, PT, PhD, Study Chair — University of Utah
Locations (1):
- Madigan Army Medical Center, Tacoma, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Any data sharing must go through a Data Sharing Agreement through the Defense Health Agency
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 3 years
Access Criteria: Any data sharing must go through a Data Sharing Agreement through the Defense Health Agency
URL: https://www.health.mil/Military-Health-Topics/Privacy-and-Civil-Liberties/Submit-a-Data-Sharing-Application

REFERENCES:
- [Background] Fritz JM, Childs JD, Wainner RS, Flynn TW. Primary care referral of patients with low back pain to physical therapy: impact on future health care utilization and costs. Spine (Phila Pa 1976). 2012 Dec 1;37(25):2114-21. doi: 10.1097/BRS.0b013e31825d32f5. PMID 22614792
- [Background] Fritz JM, Brennan GP, Hunter SJ, Magel JS. Initial management decisions after a new consultation for low back pain: implications of the usage of physical therapy for subsequent health care costs and utilization. Arch Phys Med Rehabil. 2013 May;94(5):808-16. doi: 10.1016/j.apmr.2013.01.008. Epub 2013 Jan 18. PMID 23337426
- [Background] Fritz JM, Cleland JA, Speckman M, Brennan GP, Hunter SJ. Physical therapy for acute low back pain: associations with subsequent healthcare costs. Spine (Phila Pa 1976). 2008 Jul 15;33(16):1800-5. doi: 10.1097/BRS.0b013e31817bd853. PMID 18628714
- [Derived] Rhon DI, Miller RB, Fritz JM. Effectiveness and Downstream Healthcare Utilization for Patients That Received Early Physical Therapy Versus Usual Care for Low Back Pain: A Randomized Clinical Trial. Spine (Phila Pa 1976). 2018 Oct 1;43(19):1313-1321. doi: 10.1097/BRS.0000000000002619. PMID 29489568
- [Derived] Rhon D, Fritz J. COMParative Early Treatment Effectiveness between physical therapy and usual care for low back pain (COMPETE): study protocol for a randomized controlled trial. Trials. 2015 Sep 23;16:423. doi: 10.1186/s13063-015-0959-8. PMID 26399603

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care (UC) | Early Physical Therapy (PT)
Started | 61 | 58
Completed | 61 | 58
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care (UC) | Early Physical Therapy (PT) | Total
Number analyzed (Participants) | 61 | 58 | 119
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 61 | 58 | 119
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.9 (6.3) | 29.1 (6.7) | 28.1 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 20
  Male | 49 | 50 | 99
Region of Enrollment [Number; unit: participants]
  United States | 61 | 58 | 119

OUTCOME MEASURES:

1. Primary Outcome: Modified Oswestry Disability Index
Description: The Modified Oswestry Disability Questionnaire (OSW) is a 10-item condition-specific measure of functional status (pain and disability) for patients with low back pain (LBP). Each question has 6 possible answers (0 = worse, 5 = best). The raw score is doubled to provide a percent score from 0 to 100%; with 0 equaling no disability and 100% equalling the worst possible outcome. It measures pain-related disability. We used the modified version that replaces the sex life item with an employment/ homemaking item due to poor compliance with the former. The OSW is widely used in research on non-operative management of patients with LBP, with high levels of test-retest reliability among stable patients (ICC = 0.90), good construct validity, and responsiveness to change for patients with acute LBP. It has a minimum clinically important difference of 6 points.
Time Frame: 12 months
Population: Active duty Soldiers in the United States Army
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Usual Care (UC) | Early Physical Therapy (PT)
Number analyzed (Participants) | 61 | 58
score on a scale | 23.46 [18.91 to 28.00] | 24.26 [19.82 to 28.69]

2. Secondary Outcome: Numeric Pain Rating Scale (NPRS)
Description: A 0-10 numeric pain rating scale ('0' indicating no pain, and '10' worst imaginable pain) will be used to assess LBP intensity. Numeric pain scales are known to have excellent test-retest reliability. Previous research has found the NPRS to be responsive to change, with a minimum clinically important difference of two points among patients with acute LBP receiving physical therapy.
Time Frame: 12 months
Population: Active duty Soldiers in US Army
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care (UC) | Early Physical Therapy (PT)
Number analyzed (Participants) | 58 | 55
units on a scale | 3.7 [3.0 to 4.4] | 3.7 [3.1 to 4.4]

3. Secondary Outcome: Global Rating of Change (GRC) of +3 or More (Minimum Clinically Important Change)
Description: The GRC is a 15-point scale that asks the patient to rate the degree of change in his or her condition from the beginning of treatment to the present. The mid-point of the scale is no change (0). Ratings from -1 to -7 represent varying degrees of a worsening of the patient's condition, while rating from +1 to +7 represent varying degrees of improvement. A score of 3 or higher is considered clinically meaningful change.
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care (UC) | Early Physical Therapy (PT)
Number analyzed (Participants) | 61 | 58
Participants | 16 | 20

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse events were reported to the Institutional Review Board if occurred
Arm/Group | Usual Care (UC) | Early Physical Therapy (PT)
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/58
Other Adverse Events (participants affected / at risk) | 0/61 | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No